CLINICAL TRIAL: NCT03311048
Title: Airway Inflammatory Profile Among Cleaning Workers From Different Workplaces
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Universidade Cidade de Sao Paulo (Other); Instituto de Assistencia Medica ao Servidor Publico Estadual, Sao Paulo (Other)
Responsible Party: Principal Investigator, Beatriz Mangueira Saraiva Romanholo, Clinical Professor, University of Sao Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 15149013.3.0000.5463
Record Dates: First submitted 2017-05-19; First posted 2017-10-16 (Actual); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Inflammation; Work Related Illnesses; Symptoms and Signs; Asthma, Occupational; Rhinitis
Keywords: Cleaning workers; Work-related asthma; Work-related rhinitis; Respiratory symptoms; Nasal swab
MeSH Terms: conditions — Inflammation; Signs and Symptoms; Asthma, Occupational; Rhinitis; Signs and Symptoms, Respiratory | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: : This study included 167 participants, divided in four groups based on workplace: Hospital, University, Housekeeper and Control. Nasal swab was collect to upper airways inflammation evaluation. Clinical profile and respiratory symptoms employees' evaluation were performed using specific questionnaires (European Community Respiratory Health Survey for occupational diseases evaluation (ECRHS), (adapted by Ribeiro et al, 2007) and the International Study of Asthma and Allergies in Childhood (ISAAC) - Asthma module, previously translated and validated.
Who Masked: Participant
Masking Description: Participants, divided in four groups based on workplace: Hospital, University, Housekeeper and Control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hospital (Experimental): Hospital cleaning workers Nasal swab was collect to upper airways inflammation evaluation. Clinical profile and respiratory symptoms employees' evaluation were performed using specific questionnaires (European Community Respiratory Health Survey for occupational diseases evaluation (ECRHS), (adapted by Ribeiro et al, 2007) and the International Study of Asthma and Allergies in Childhood (ISAAC) - Asthma module, previously translated and validated.
  Interventions: Other: Nasal swab; Other: Questionnaires
- University (Experimental): Campus (university) cleaning workers Nasal swab was collect to upper airways inflammation evaluation. Clinical profile and respiratory symptoms employees' evaluation were performed using specific questionnaires (European Community Respiratory Health Survey for occupational diseases evaluation (ECRHS), (adapted by Ribeiro et al, 2007) and the International Study of Asthma and Allergies in Childhood (ISAAC) - Asthma module, previously translated and validated.
  Interventions: Other: Nasal swab; Other: Questionnaires
- Housekeeper (Experimental): Housemaid (cleaning workers) Nasal swab was collect to upper airways inflammation evaluation. Clinical profile and respiratory symptoms employees' evaluation were performed using specific questionnaires (European Community Respiratory Health Survey for occupational diseases evaluation (ECRHS), (adapted by Ribeiro et al, 2007) and the International Study of Asthma and Allergies in Childhood (ISAAC) - Asthma module, previously translated and validated.
  Interventions: Other: Nasal swab; Other: Questionnaires
- Control (Experimental): Office workers (no relationship to cleaning) Nasal swab was collect to upper airways inflammation evaluation. Clinical profile and respiratory symptoms employees' evaluation were performed using specific questionnaires (European Community Respiratory Health Survey for occupational diseases evaluation (ECRHS), (adapted by Ribeiro et al, 2007) and the International Study of Asthma and Allergies in Childhood (ISAAC) - Asthma module, previously translated and validated.
  Interventions: Other: Nasal swab; Other: Questionnaires

INTERVENTIONS:
Other: Nasal swab — Nasal swab was collect to upper airways inflammation evaluation.
Other: Questionnaires — Clinical profile and respiratory symptoms employees' evaluation were performed using specific questionnaires (European Community Respiratory Health Survey for occupational diseases evaluation (ECRHS), (adapted by Ribeiro et al, 2007) and the International Study of Asthma and Allergies in Childhood (ISAAC) - Asthma module, previously translated and validated.

SUMMARY:
There are consistent evidences through epidemiologic studies in different places, reinforced by occupational asthma records studies, that cleaning workers have a high risk in developing asthma. These risk determinants are not totally known. The air around the worker may have some higher and lower molecular weight with different concentration peaks from removed dust of the cleaning process and volatile substances from cleaning products. Cleaning activities may occur in different places. Although the relationship between rhinitis and asthma is already established, there are not many studies about occupational rhinitis-related work place. This study aimed to investigate airway inflammation and respiratory symptoms of cleaning workers from different workplaces.

DETAILED DESCRIPTION:
Were recruited to participate in the study individuals from four different workplaces: Hospital; University; Housekeeper and Control (office workers). The research was performed in Cacoal city, Rondonia, Brazil. Smokers (active), pregnant, lactating, and individuals at continuing therapy for treating disorders of the airways were excluded.

Clinical profile and respiratory symptoms employees evaluation were performed using the European Community Respiratory Health Survey for occupational diseases evaluation (ECRHS), and the International Study of Asthma and Allergies in Childhood (ISAAC) - Asthma module.

Nasal swab was collected for evaluation of upper airways inflammation, according to Ronchetti et al protocol, using a sterile swab that was moistened with 1mL saline solution; both nostrils were scraped using this swab. Twenty minutes after this, laminas were stained using May-Grunwald-Giemsa to eosinophils, neutrophils, lymphocytes, macrophages and epithelial cells identification. Cells were analyzed using a Nikon E600 optical microscope (Nikon, Canada), of 1.000 x magnitude. Whenever possible a total of 200 cells were counted in two slides.

Statistical analysis were performed using Anova variance (Kruskal-Wallis) and Dunn's test for comparisons between groups. To evaluate the association between the qualitative variables we used the chi-square, Statistical software Sigma Plot 12.0 and SPSS 21.0. The confidence interval was 95% (p <0.05).

ELIGIBILITY:
Inclusion Criteria:

* Cleaning workers from different workplaces
* Non-cleaning workers (control group)
* People legally capable (over 18 years old)
* Must be able to nasal swab collection and answer questionnaires
* Sign the informed consent form

Exclusion Criteria:

* Smokers (active)
* Pregnant (women)
* Lactating (women)
* Not accept the informed consent form
* Individuals at continuing therapy for airways treating disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Measure of respiratory symptoms | One day
  Questionnaires to analyze respiratory symptons
Cell differentiation for the evaluation of nasal epithelial inflammation | One day
  Nasal swab will be collected to analyze cell differentiation

CONTACTS AND LOCATIONS:
Overall Officials: BEATRIZ BS Mangueira Saraiva-Romanholo, PhD, Study Chair — Universidade Cidade de Sao Paulo; Edineia R Paz, Master, Study Chair — Instituto de Assistencia Medica ao Servidor Publico Estadual, Sao Paulo
Locations (1):
- Children's Institute of the Clinical Hospital of University of Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ocansey S, Tatton-Brown K. EZH2-Related Overgrowth. 2013 Jul 18 [updated 2025 Jun 26]. In: Adam MP, Bick S, Mirzaa GM, Pagon RA, Wallace SE, Amemiya A, editors. GeneReviews(R) [Internet]. Seattle (WA): University of Washington, Seattle; 1993-2026. Available from http://www.ncbi.nlm.nih.gov/books/NBK148820/ PMID 23865096
- [Background] Aun MV, Saraiva-Romanholo BM, Almeida FM, Bruggemann TR, Kalil J, Martins Mde A, Arantes-Costa FM, Giavina-Bianchi P. Sensitization by subcutaneous route is superior to intraperitoneal route in induction of asthma by house dust mite in a murine mode. Einstein (Sao Paulo). 2015 Oct-Dec;13(4):560-6. doi: 10.1590/S1679-45082015AO3389. PMID 26761554
- [Background] da Silva RA, Almeida FM, Olivo CR, Saraiva-Romanholo BM, Perini A, Martins MA, Carvalho CR. Comparison of the effects of aerobic conditioning before and after pulmonary allergic inflammation. Inflammation. 2015;38(3):1229-38. doi: 10.1007/s10753-014-0090-0. PMID 25537797
- [Background] Brito JM, Macchione M, Yoshizaki K, Toledo-Arruda AC, Saraiva-Romanholo BM, Andrade Mde F, Mauad T, Rivero DH, Saldiva PH. Acute cardiopulmonary effects induced by the inhalation of concentrated ambient particles during seasonal variation in the city of Sao Paulo. J Appl Physiol (1985). 2014 Sep 1;117(5):492-9. doi: 10.1152/japplphysiol.00156.2014. Epub 2014 Jul 10. PMID 25012028
- [Background] Possa SS, Charafeddine HT, Righetti RF, da Silva PA, Almeida-Reis R, Saraiva-Romanholo BM, Perini A, Prado CM, Leick-Maldonado EA, Martins MA, Tiberio Ide F. Rho-kinase inhibition attenuates airway responsiveness, inflammation, matrix remodeling, and oxidative stress activation induced by chronic inflammation. Am J Physiol Lung Cell Mol Physiol. 2012 Dec 1;303(11):L939-52. doi: 10.1152/ajplung.00034.2012. Epub 2012 Sep 21. PMID 23002076
- [Background] Manzano RM, Carvalho CR, Saraiva-Romanholo BM, Vieira JE. Chest physiotherapy during immediate postoperative period among patients undergoing upper abdominal surgery: randomized clinical trial. Sao Paulo Med J. 2008 Sep;126(5):269-73. doi: 10.1590/s1516-31802008000500005. PMID 19099160
- [Background] de Amorim CG, Sa Malbouisson LM, Saraiva BM, Pedro FM, Martins MA, Carmona MJ. Evaluation of exhaled nitric oxide in patients undergoing myocardial revascularization with cardiopulmonary bypass. Rev Bras Anestesiol. 2009 May-Jun;59(3):286-96. doi: 10.1590/s0034-70942009000300003. English, Portuguese. PMID 19488541
- [Background] Saraiva-Romanholo BM, Barnabe V, Carvalho AL, Martins MA, Saldiva PH, Nunes Mdo P. Comparison of three methods for differential cell count in induced sputum. Chest. 2003 Sep;124(3):1060-6. doi: 10.1378/chest.124.3.1060. PMID 12970038
- [Background] Palomino AL, Bussamra MH, Saraiva-Romanholo BM, Martins MA, Nunes Mdo P, Rodrigues JC. [Induced sputum in children and adolescents with asthma: safety, clinical applicability and inflammatory cells aspects in stable patients and during exacerbation]. J Pediatr (Rio J). 2005 May-Jun;81(3):216-24. Portuguese. PMID 15951906
- [Background] Paro-Heitor ML, Bussamra MH, Saraiva-Romanholo BM, Martins MA, Okay TS, Rodrigues JC. Exhaled nitric oxide for monitoring childhood asthma inflammation compared to sputum analysis, serum interleukins and pulmonary function. Pediatr Pulmonol. 2008 Feb;43(2):134-41. doi: 10.1002/ppul.20747. PMID 18085692
- [Background] Saraiva-Romanholo BM, Machado FS, Almeida FM, Nunes Mdo P, Martins MA, Vieira JE. Non-asthmatic patients show increased exhaled nitric oxide concentrations. Clinics (Sao Paulo). 2009;64(1):5-10. doi: 10.1590/s1807-59322009000100002. PMID 19142544
- [Background] Mendes FA, Goncalves RC, Nunes MP, Saraiva-Romanholo BM, Cukier A, Stelmach R, Jacob-Filho W, Martins MA, Carvalho CR. Effects of aerobic training on psychosocial morbidity and symptoms in patients with asthma: a randomized clinical trial. Chest. 2010 Aug;138(2):331-7. doi: 10.1378/chest.09-2389. Epub 2010 Apr 2. PMID 20363839
- [Background] Hizume DC, Toledo AC, Moriya HT, Saraiva-Romanholo BM, Almeida FM, Arantes-Costa FM, Vieira RP, Dolhnikoff M, Kasahara DI, Martins MA. Cigarette smoke dissociates inflammation and lung remodeling in OVA-sensitized and challenged mice. Respir Physiol Neurobiol. 2012 Apr 30;181(2):167-76. doi: 10.1016/j.resp.2012.03.005. Epub 2012 Mar 15. PMID 22446562
- [Background] Silva RA, Almeida FM, Olivo CR, Saraiva-Romanholo BM, Martins MA, Carvalho CR. Exercise reverses OVA-induced inhibition of glucocorticoid receptor and increases anti-inflammatory cytokines in asthma. Scand J Med Sci Sports. 2016 Jan;26(1):82-92. doi: 10.1111/sms.12411. Epub 2015 Feb 4. PMID 25652754
- [Derived] da Paz ER, de Lima CMF, Felix SN, Schaeffer B, Galvao CES, Correia AT, Righetti RF, de Arruda Martins M, de Fatima Lopes Calvo Tiberio I, Saraiva-Romanholo BM. Airway inflammatory profile among cleaning workers from different workplaces. BMC Pulm Med. 2022 Apr 29;22(1):170. doi: 10.1186/s12890-022-01949-5. PMID 35488256
- Available data/document: Informed Consent Form: Sistema Nacional de Informação — http://portal2.saude.gov.br/sisnep/pesquisador